CLINICAL TRIAL: NCT05426486
Title: A Randomized, Open Label, Multi-center Phase II-III Neoadjuvant Study Comparing the Efficacy and Safety of ARX788 Combined With Pyrotinib Maleate Versus TCBHP (Trastuzumab Plus Pertuzumab With Docetaxel and Carboplatin) in Patients With HER2-positive Breast Cancer
Brief Title: A Study of ARX788 Combined With Pyrotinib Maleate Versus TCBHP (Trastuzumab Plus Pertuzumab With Docetaxel and Carboplatin) as Neoadjuvant Treatment in HER2-positive Breast Cancer Patients
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Caigang Liu (Other)
Responsible Party: Sponsor-Investigator, Caigang Liu, Director of the Cancer Center, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUKDEN 06
Record Dates: First submitted 2022-06-12; First posted 2022-06-22 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: HER2-positive Breast Cancer
Keywords: ARX788; Pyrotinib; HER2-positive Breast Cancer; Neoadjuvant
MeSH Terms: interventions — ARX788; Trastuzumab; pertuzumab; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARX788 + pyrotinib maleate (Experimental): ARX788 1.5 mg/kg intravenously (IV) every three weeks plus pyrotinib maleate 320 mg orally once daily for 6 cycles
  Interventions: Drug: ARX788; Drug: Pyrotinib maleate
- trastuzumab + pertuzumab + docetaxel + carboplatin (Active Comparator): Trastuzumab (8 mg/kg first dose, followed 6 mg/kg) puls pertuzumab (840 mg first dose, followed 420 mg) plus docetaxel (75 mg/m3) plus carboplatin (AUC6) IV every 3 weeks for 6 cycles
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Docetaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: ARX788 — HER2 antibody-drug conjugate
  Arms: ARX788 + pyrotinib maleate
Drug: Pyrotinib maleate — EGFR/HER2 dual inhibitor
  Arms: ARX788 + pyrotinib maleate
Drug: Trastuzumab — anti-Her2 monoclonal antibody
  Arms: trastuzumab + pertuzumab + docetaxel + carboplatin
Drug: Pertuzumab — anti-HER2 monoclonal antibody
  Arms: trastuzumab + pertuzumab + docetaxel + carboplatin
Drug: Docetaxel — Cytotoxic chemotherapy
  Arms: trastuzumab + pertuzumab + docetaxel + carboplatin
Drug: Carboplatin — Cytotoxic chemotherapy
  Arms: trastuzumab + pertuzumab + docetaxel + carboplatin

SUMMARY:
This is a randomized, open label Phase II-III neoadjuvant study comparing the efficacy and safety of ARX788 combined with pyrotinib maleate versus TCBHP (trastuzumab plus pertuzumab with docetaxel and carboplatin) in patients with HER2-positive breast cancer.

DETAILED DESCRIPTION:
This is a randomized, open label Phase II-III neoadjuvant study comparing the efficacy and safety of ARX788 combined with pyrotinib maleate versus TCBHP (trastuzumab plus pertuzumab with docetaxel and carboplatin) in patients with HER2-positive breast cancer. Patients will be randomized (1:1) to one of the two treatment arms: arm 1, ARX788 plus pyrotinib maleate for 6 cycles; arm 2, trastuzumab plus pertuzumab with docetaxel and carboplatin for six cycles. Patients will undergo surgery after neoadjuvant therapy. Efficacy will be assessed every 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 but ≤ 75 years;
* Diagnosis of breast cancer meets the following criteria: Histologically confirmed invasive breast cancer; Tumor staging: Stage II-III patients who meet the 8th edition of AJCC Cancer Staging Manual;
* HER2-positive breast cancer pathologically confirmed is defined as Immunohistochemical method (IHC 3+) or IHC 2+ with FISH+;
* Eastern Cooperative Oncology Group (ECOG) level 0-1;
* The functional level of major organs must conform to the following requirements: Neutrophils (ANC) ≥ 1.5×10^9/L (with no use of growth factors within 14 days); Platelet count (PLT) ≥ 100×10^9/L (with no correct treatment within 7 days ); Hemoglobin (Hb) ≥ 90 g/L (with no correct treatment within 7 days ); Total bilirubin (TBIL) ≤ 1.5×upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3×ULN; Urea nitrogen and creatinine ≤ 1.5×ULN and creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula); Cardiac color Doppler ultrasound: left ventricular ejection fraction (LVEF) ≥ 50%; 12-lead electrocardiogram: QT interval ≤ 480 ms;
* Patients who participate in the trial voluntarily, sign an informed consent, have good compliance and are willing to comply with the follow-up visit.

Exclusion Criteria:

* Previously received any anti-tumor therapy (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.);
* Patients who are concurrently receiving other anti-tumor therapy;
* Bilateral breast cancer, inflammatory breast cancer, or occult breast cancer;
* Stage IV breast cancer;
* With a history of any malignancies other than breast cancer in the past 5 years, excluding cured cervical carcinoma in situ and melanoma skin cancer;
* Inability to swallow, chronic diarrhea and intestinal obstruction, and having many factors that affect drug administration and absorption;
* Patients with known allergies to any active ingredients or excipients of Investigational medicinal product;
* With a history of interstitial pulmonary disease, drug-induced pulmonary interstitial disease, and radiation pneumonitis that require hormone therapy, or any clinically active pulmonary interstitial disease as suggested by any evidence;
* Patients who are currently suffering from keratitis, corneal disease, retinal disease, or active eye infection that require any interventions for the eyes;
* Once suffered from any heart disease, including: (1) arrhythmia with clinical significance, (2) myocardial infarction; (3) heart failure; (4) investigator's judgment as not suitable for participating in this trial;
* Female patients during pregnancy and lactation, or those who are fertile and positive for baseline pregnancy test or those of childbearing age who are unwilling to take effective contraceptive measures throughout the trial period;
* Serious concomitant diseases or other comorbid diseases that will endanger the safety of patients or interfere with the completion of the trial, including but not limited to severe hypertension, severe diabetes mellitus, and active infections that are out of control;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Total pathological complete response rate (tpCR) rate | 3 years
  The standard for removal of breast and lymph node tumors which means there are no infiltrating cancer cells at the primary breast and axillary lymph nodes, and only intraductal cancer is allowed on the breast.

SECONDARY OUTCOMES:
Breast pathological complete response rate (bpCR) rate | 3 years
  The standard for breast tumor removal which means that there are only infiltrating cancer cells at the primary breast tumor site.
Residual tumor burden (RCB) | 3 years
  Postoperative pathological results will be used to assess the residual tumor area of primary breast tumor (area in mm×mm), the cell density of the residual tumor（cell density in percentages）, the proportion of carcinoma in situ (proportion of carcinoma in percentages), the number of positive lymph nodes and the diameter of largest metastasis with residual nodes (diameter in mm). The RCB class can be estimated from the above five pathological parameters through a network calculation: RCB-0 in grades: pCR; RCB-I in grades: minimal residual tumor; RCB-II: moderate residual tumor; RCB-III in grades: extensive residual tumor.
Best overall response rate (BORR) | 3 years
  The proportion of patients who achieve remission at any point during the study.
Five-year overall survival (OS) | 5 years
  The time from the random date to death due to any cause.
Event-free survival (EFS) | 3 years
  The time from the day of enrollment to the first occurrence of recurrent disease, including second primary malignancies in the non-breast area and breast ductal carcinoma in situ.
Adverse events (AE) | 3 years
  Adverse events (AE) will be assessed as per the NCI-CTC AE 5.0 standard.

CONTACTS AND LOCATIONS:
Overall Officials: Caigang Liu, MD, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No